CLINICAL TRIAL: NCT06577389
Title: Enhanced Recovery After Surgery for Spine Fusion Surgeries in the Elderly
Acronym: ERAS in Spine
Status: Not yet recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Aikeremujiang Muheremu, MD,PhD, Sixth Affiliated Hospital of Xinjiang Medical University
Other Study IDs: SixthAHXinjiang
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Spinal Stenosis
Keywords: spine fusion surgery
MeSH Terms: conditions — Spinal Stenosis | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly after spine fusion surgery: patients receive Enhanced recovery after spinal fusion surgery
  Interventions: Other: Enhanced recovery after surgery

INTERVENTIONS:
Other: Enhanced recovery after surgery — The ERAS program for lumbar fusion surgery will be implemented.

SUMMARY:
elderly patients in our hospital who received spinal fusion surgery after the year 2025 will receive ERAS treatment.

ELIGIBILITY:
Inclusion Criteria:

* elderly patients who received spinal fusion surgeries

Exclusion Criteria:

* patients who received non-fusion surgeries

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly patients who received spinal fusion surgeries
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
ambulation time | 7 days

SECONDARY OUTCOMES:
mean hospital length of stay | one month
cost of hosptial stay | 1 months

IPD SHARING:
Plan to Share IPD: Undecided
will decide before the year 2026